CLINICAL TRIAL: NCT01162252
Title: Improving Psoriasis Through Health and Well-Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jan Moynihan, Director, The Rochester Center for Mind-Body Research, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01AT005082 (NIH); R01AT005082-01A1 (NIH)
Record Dates: First submitted 2010-06-21; First posted 2010-07-14 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Psoriasis
Keywords: psoriasis; mindfulness; MBSR; stress; living well
MeSH Terms: conditions — Psoriasis | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness-Based Stress Reduction (Active Comparator)
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Living Well (Active Comparator)
  Interventions: Behavioral: Living Well

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — The standardized Mindfulness-Based Stress Reduction (MBSR) program is the primary training tool used to enhance mindfulness. The eight-week-long MBSR program is designed to teach subjects how to develop their inner resources in the service of taking better care of themselves. MBSR training includes the learning and refining of a range of skills aimed at increasing relaxation and awareness of physical experiences and sensations related to physical symptoms, emotions, and thoughts. Special emphasis is placed on movement, meditation, and breathing.
  Other Names: MBSR
  Arms: Mindfulness-Based Stress Reduction
Behavioral: Living Well — The Living Well (LW) program involves a series of informational presentations and group discussions on a variety of topics related to the promotion of health and well-being. The 8-week program is designed to provide participants with knowledge about ways to improve their physical and emotional health as a complement to traditional medical treatments.
  Other Names: LW
  Arms: Living Well

SUMMARY:
The purpose of the study is to examine and compare the effects of the Mindfulness-Based Stress Reduction (MBSR) program and the Living Well (LW) program on adults with psoriasis in terms of how these programs may affect their psoriasis, immune function, physical and emotional health, and well-being.

DETAILED DESCRIPTION:
The study examines the effects of two eight-week programs (MBSR vs. LW) for disease processes in patients with psoriasis severity reporting moderate or higher perceived stress. The research will focus both on clinical measures of the disease state and overall well-being.

The Aims of our proposed intervention study are the following:

1. To examine the effects of MBSR, versus the Living Well (LW) program, on (a) disease severity, immunological markers of inflammation, and keratinocyte proliferation, (b) psoriasis-related stress and perceived stress in general, and (c) anxiety and depression.
2. To examine whether treatment effects of either program are moderated by personality traits, mindfulness, and age.
3. To examine the effects of behavioral and psychological mediators on immune outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* English speaking
* Clinical diagnosis of psoriasis (active at initial visit)

Exclusion Criteria:

* currently receiving immunosuppressive therapy for cancer or for diseases unrelated to psoriasis (or < 6 months post-chemo or radiation)
* major, uncorrected sensory impairments
* cognitive deficits (MMSE <25, or deficits deemed significant enough to interfere)
* severe cardiovascular disease
* current alcohol abuse or non-alcohol psychoactive substance use disorders, psychotic disorders (current and lifetime), and current mood disorder with psychotic features.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Psoriasis disease severity measured from biopsied tissue samples of psoriatic and nonpsoriatic skin. | 8 weeks
  Psoriasis is assessed for keratinocyte proliferation including immunohistochemistry (for CD3, neutrophil elastase, keratin 6 and S100A7 markers) and quantitative real time polymerase chain reaction (qRT-PCR) to examine expression of mRNA for IFN-γ, TNF-α, IL-17A, and the shared p40 subunit of IL-12 and IL-23 (assessed pre & post intervention).

SECONDARY OUTCOMES:
Immunological markers of inflammation measured from blood samples. | 16 weeks
  Circulating cytokines IL-6, TNF-α, and IL-22 measured via enzyme-linked immunoassays (ELISA) on all blood samples (pre, mid & post intervention plus follow-up).
Perceived Stress Scale (Cohen S., Kamarck T., & Mermelstein R. (1983)) | 16 weeks
  The 14-item Perceived Stress Scale (PSS) is used to measure the degree to which current life situations are appraised as stressful by a participant (assessed at pre, mid & post intervention plus follow-up).
State-Trait Anxiety Inventory (Spielberger C.D., Gorsuch R.L., & Lushene R.E. (1970)) | 16 weeks
  The State-Trait Anxiety Inventory (STAI) consists of two, 20-item scales to distinguish between relatively recent, transitory "state anxieties", from more chronic or persistent "trait anxiety" (assessed pre, mid & post intervention plus follow-up).

CONTACTS AND LOCATIONS:
Overall Officials: Jan A Moynihan, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester; University Dermatology Associates, Rochester, New York, United States

REFERENCES:
- See also: The Rochester Center for Mind-Body Research (RCMBR) — http://www.urmc.rochester.edu/psychiatry/research/rcmbr/index.cfm
- See also: Psoriasis Center (University of Rochester Medical Center) — http://www.urmc.rochester.edu/dermatology/psoriasis